CLINICAL TRIAL: NCT01855126
Title: Individually Tailored Lighting System to Improve Sleep in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rensselaer Polytechnic Institute (Other)
Collaborators: University of North Carolina (Other)
Responsible Party: Principal Investigator, Mariana G Figueiro, Professor, Rensselaer Polytechnic Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AG042602 (NIH)
Record Dates: First submitted 2013-05-09; First posted 2013-05-16 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Sleep Disturbances
Keywords: light; circadian rhythms; dim light melatonin onset; sleep
MeSH Terms: conditions — Parasomnias | interventions — Blue Light; Red Light

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized to receive either the active intervention or placebo intervention and then crossed over to receive the opposite intervention. The study consisted of two intervention periods of 8 weeks separated by a two week washout period.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blue light (Experimental): The study protocol consisted of two 8-week intervention/control periods in which each participant wore either the intervention (blue light) or control (red light) mask every night, with the order of presentation of the two conditions randomized by the study's biostatistician. A light mask housing two blue Light Emitting Diodes (LED) arrays delivered a train of blue or red light pulses of 2 second duration that were presented every 30 s for no longer than 2 hr, resulting in a maximum total of approximately 240 pulses per night. the blue light mask was worn nightly for 8 weeks. There will be a two week washout period between each intervention
  Interventions: Other: Blue light
- Red light (Placebo Comparator): The study protocol consisted of two 8-week intervention/control periods in which each participant wore either the intervention (blue light) or control (red light) mask every night, with the order of presentation of the two conditions randomized by the study's biostatistician. A light mask housing two red Light Emitting Diodes (LED) arrays delivered a train of blue or red light pulses of 2 second duration that were presented every 30 s for no longer than 2 hr, resulting in a maximum total of approximately 240 pulses per night. the red light mask was worn nightly for 8 weeks, with a two week washout period between each intervention
  Interventions: Other: Red light

INTERVENTIONS:
Other: Blue light — After a two week baseline collection period, half of the subjects will initially be given light masks that deliver blue light through the closed eyelids, while subjects are sleeping. The light mask will always be turned on 120 min before estimated core body temperature minimum (CBTmin); it is expected that blue light exposure will delay the timing of the CBTmin.
  Arms: Blue light
Other: Red light — After a two week baseline collection period, half of the subjects will initially be given light masks that deliver red light through the closed eyelids, while subjects are sleeping. The light mask will always be turned on 120 min before estimated core body temperature minimum (CBTmin); it is expected that red light exposure will have no effect on the timing of the CBTmin.
  Arms: Red light

SUMMARY:
In conjunction with investigators at the Cecil G. Sheps Center for Health Services Research, University of North Carolina (UNC) at Chapel Hill, we propose to develop and evaluate a low-cost, minimally obtrusive device that delivers individualized light therapy to adults with early-awakening insomnia - the most common sleep disturbance in older adults, and a significant problem because of its relationship to daytime sleepiness, use of potentially hazardous sleep medication, and reduced quality of life. The proposed device will measure light/dark exposure data over 24 hours, estimate optimum timing for light delivery, and deliver an individualized light dosage while subjects are asleep. Light applied through closed eyelids in the early part of the night will delay the dim light melatonin onset, a marker of the circadian clock, and help those with early sleep onset to fall asleep later

DETAILED DESCRIPTION:
We will recruit 50 subjects who report going to bed early and desiring later bedtimes and will ask them to wear an active and an inactive light mask for 8 consecutive weeks each. A 2-week washout period between active and inactive conditions will be applied. Outcome measures will be collected periodically throughout the 8 weeks. Baseline (no intervention) will be collected prior to the active and inactive lighting interventions.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older
* cognitively capable
* able to respond to study staff verbally and in English
* score greater than 6 using the Pittsburgh Sleepiness Quality Index
* suffer from insomnia
* suffer from excessive daytime sleepiness

Exclusion Criteria:

* Severe sleep apnea
* Severe restless leg syndrome (RLS)
* Significant cognitive impairment
* History of severe photosensitivity dermatitis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana G Figueiro, PhD, Principal Investigator — Rensselaer Polytechnic Institute
Locations (1):
- Rensselaer Polytechnic Institute, Troy, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Figueiro MG, Plitnick B, Rea MS. Pulsing blue light through closed eyelids: effects on acute melatonin suppression and phase shifting of dim light melatonin onset. Nat Sci Sleep. 2014 Dec 2;6:149-56. doi: 10.2147/NSS.S73856. eCollection 2014. PMID 25506253
- [Background] Figueiro MG, Bierman A, Rea MS. A train of blue light pulses delivered through closed eyelids suppresses melatonin and phase shifts the human circadian system. Nat Sci Sleep. 2013 Oct 4;5:133-41. doi: 10.2147/NSS.S52203. eCollection 2013. PMID 24124400

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 participants were enrolled into the study. These participants were randomized to begin the study with the active intervention, or the placebo intervention. After a 2 week washout period, participants were exposed to the opposite intervention.
Groups:
- Active Intervention, Then Placebo: Participants started the study wearing the blue mask for 8 weeks. After a 2 week washout period, they wore the red mask for 8 weeks
- Placebo Intervention, Then Active: Participants started the study wearing the red mask every night for 8 weeks. After a 2 week washout period, they wore the blue mask every night for 8 weeks.
Period: First Intervention (8 Weeks)
Arm/Group | Active Intervention, Then Placebo | Placebo Intervention, Then Active
Started | 24 | 22
Completed | 20 | 16
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 4 | 6
Period: Washout Period (2 Weeks)
Arm/Group | Active Intervention, Then Placebo | Placebo Intervention, Then Active
Started | 20 | 16
Completed | 20 | 16
Not Completed | 0 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Active Intervention, Then Placebo | Placebo Intervention, Then Active
Started | 20 | 16
Completed | 18 | 14
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active Intervention, Then Placebo Intervention: Participants started the study by wearing the blue mask every night for 8 weeks. After a washout period of 2 weeks, participants wore the red mask every night for 8 weeks
- Placebo Intervention, Then Active Intervention: Participants started the study by wearing the red mask every night for 8 weeks. After a washout period of 2 weeks, participants wore the blue mask every night for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Active Intervention, Then Placebo Intervention | Placebo Intervention, Then Active Intervention | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 17 | 15 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50
early awakening insomnia [Count of Participants; unit: Participants] | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Sleep Disturbance
Description: Pittsburgh Sleep Quality Index. Score range 0 - 21. A score over 5 is indicative of sleep disturbance.
  Change in score from baseline to intervention is reported. A larger difference indicates a better outcome.
Time Frame: Baseline (week 0) and week 8 of lighting intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Blue Light Mask: Participants wore the blue mask every night for 8 weeks.
- Red Light Mask: Participants wore the red mask every night for 8 weeks.
Arm/Group | Blue Light Mask | Red Light Mask
Number analyzed (Participants) | 34 | 34
units on a scale | -1.9 (0.5) | -1.3 (0.5)

2. Primary Outcome: Total Sleep Time
Description: The change in total amount of minutes spent sleeping at night from baseline week to the last week of intervention. A higher number is an improved outcome
Time Frame: baseline week (week 0) and the last week of intervention (week 8)
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Blue Light Mask: Participants started the study wearing the blue light mask every night for 8 weeks.
- Red Light Mask: Participants started the study wearing the red light mask for 8 weeks.
Arm/Group | Blue Light Mask | Red Light Mask
Number analyzed (Participants) | 34 | 34
minutes | 4 (22) | 1 (19)

3. Primary Outcome: Sleep Efficiency
Description: The change in sleep efficiency from baseline to last week of intervention. A higher number is a better outcome. Sleep efficiency is the percentage of time spent in bed sleeping. Scored total sleep time divided by interval duration minus total invalid time (sleep/wake) of the given rest interval multiplied by 100. This data was collected using actigraphy data.
Time Frame: baseline week (week 0) and the last week of intervention (week 8)
Measure: Mean (Standard Deviation); unit: percentage of sleep
Groups:
- Blue Light Mask: Participants started the study wearing the blue mask for 8 weeks.
- Red Light Mask: Participants started the study wearing the red mask every night for 8 weeks.
Arm/Group | Blue Light Mask | Red Light Mask
Number analyzed (Participants) | 34 | 34
percentage of sleep | 1.3 (2.9) | -0.6 (4.7)

4. Primary Outcome: Sleep Start Time
Description: Change in sleep start time, in minutes, from baseline week to the last week of intervention. A higher number is a better outcome. Based on actigraph data
Time Frame: baseline week (week 0) and the last week of intervention (week 8)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Blue Light Mask | Red Light Mask
Number analyzed (Participants) | 34 | 34
minutes | 9 (21) | 1 (3)

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: data was collected weekly during each 8 week intervention period
Groups:
- Blue Light: This within-subjects, randomized, two-treatment crossover design study consists of two 8-week periods in which each participant wore either the intervention (blue light) or control (red light) mask every night. Subjects will use each condition for eight weeks, with the intervention order counterbalanced across subjects, and a two-week washout period between the two study conditions. The blue mask delivered a flashing blue light for two hours beginning 1 hour after bedtime designed to result in a phase delay of the circadian response curve.
- Red Light: This within-subjects, randomized, two-treatment crossover design study consists of two 8-week periods in which each participant wore either the intervention (blue light) or control (red light) mask every night. Subjects will use each condition for eight weeks, with the intervention order counterbalanced across subjects, and a two-week washout period between the two study conditions. The red mask delivered a flashing red light for two hours beginning 1 hour after bedtime designed to have no effect on the circadian response curve.
Arm/Group | Blue Light | Red Light
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 13/34 | 12/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blue Light (N=34) | Red Light (N=34)
Eye Burning (Eye disorders) | 13 | 12
Eye Redness (Eye disorders) | 10 | 10
Eye strain (Eye disorders) | 9 | 8
Headache (General disorders) | 13 | 12

LIMITATIONS AND CAVEATS:
We did not collect circadian marker data (e.g., DLMO) in this field study, it is not known whether any circadian phase shifting resulted. We did not control light during the day which could have counteracted the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT01855126/SAP_000.pdf
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT01855126/Prot_001.pdf